CLINICAL TRIAL: NCT07149623
Title: A Prospective Multicenter Observational Study on Metastatic Lymph Node Distribution of Ileum Mesentery in Cecal Cancer and Proximal Ascending Colon Cancer
Brief Title: Metastatic Lymph Node Distribution in the Ileum Mesentery of Cecal and Proximal Ascending Colon Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, XIAO Yi, MD, XIAO Yi, Peking Union Medical College Hospital
Other Study IDs: RELARC-02
Record Dates: First submitted 2025-07-21; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-07

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- experimental group
  Interventions: Procedure: Experimental

INTERVENTIONS:
Procedure: Experimental — sectioning and submitting fresh surgical specimens from the ileum mesentery

SUMMARY:
Based on the above considerations, our team maintains that it is currently imperative to conduct a prospective multicenter registry study. This study would involve sectioning and submitting fresh surgical specimens from the ileum mesentery of patients undergoing radical resection for cecal cancer and proximal ascending colon cancer (right-sided colon cancer). The objectives are to: Clarify the distribution range of metastatic lymph nodes within the ileum mesentery; Conduct survival follow-up on enrolled patients; Provide reliable evidence-based medical evidence for the individualized determination of ileal resection margins.

ELIGIBILITY:
Inclusion Criteria:

Age 18-80 years; ECOG performance status 0-2; Histologically confirmed colon adenocarcinoma; Surgical specimen confirming tumor location at: ileocecal valve orifice (cecal cancer), OR proximal ascending colon cancer with tumor ≤5 cm from ileocecal valve; Clinical stage: cT2-4aN0M0, OR cTanyN+M0; Patient and family members fully understand the study and voluntarily participate by signing informed consent

Exclusion Criteria:

Synchronous or metachronous multiple primary colon cancers (Note: Synchronous: diagnosed within 6 months; Metachronous: diagnosed >6 months apart); Preoperative neoadjuvant therapy (chemotherapy, immunotherapy, or radiotherapy) that may cause tumor regression or downstaging; Patients undergoing salvage radical surgery after endoscopic resection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with cecal cancer and proximal ascending colon cancer
Sampling Method: Non-Probability Sample
Enrollment: 406 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Metastatic rate in mesenteric lymph nodes | 1 month after surgery

SECONDARY OUTCOMES:
Distribution of metastatic lymph nodes in the mesentery | 1 month after surgery
3-year disease-free survival | 3 years after surgery
5-year overall survival | 5 years after surgery

IPD SHARING:
Plan to Share IPD: No